CLINICAL TRIAL: NCT00873665
Title: Exercise Training, Erectile Dysfunction, and Prostate Cancer Study.
Brief Title: Erectile Dysfunction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011329; CA133895-01
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): To determine the effects of supervised aerobic exercise training versus usual care on incidence of ED among men undergoing radical prostatectomy for clinically localized prostate cancer.
  The test of the arm effect of incidence of ED will be made with the Wald chi-square test from the logistic regression model. A dichotomous variable indicating whether the patient received PDE-5 inhibitor therapy will be used as a covariate in the model. The arm effect will be summarized by giving arm-specific covariate-adjusted proportions and their 80% confidence intervals, and the p-value.
  Interventions: Other: aerobic exercise
- Wait-list control (Other): To determine the effects of aerobic exercise training versus wait-list control on changes in patient symptoms (i.e., erectile function score, sexual functioning, urinary incontinence, and QOL) and the number of men receiving phosphodiesterases type-5 (PDE-5) inhibitor therapy as well as therapy dose.
  For the analyses of arm differences in erectile dysfunction (IIEF) score, sexual functioning, urinary incontinence, and QOL, the primary endpoints will be the change across time in these continuous variables. Specifically, change across time for LTF patients will be imputed to be zero for all these analyses.
  Interventions: Other: wait-list control

INTERVENTIONS:
Other: aerobic exercise — To determine the effects of supervised aerobic exercise training versus usual care on incidence of ED among men undergoing radical prostatectomy for clinically localized prostate cancer.
  Other Names: Erectile Dysfunction
  Arms: Aerobic exercise
Other: wait-list control — To determine the effects of aerobic exercise training versus wait-list control on changes in patient symptoms (i.e., erectile function score, sexual functioning, urinary incontinence, and QOL) and the number of men receiving phosphodiesterases type-5 (PDE-5) inhibitor therapy as well as therapy dose.
  Other Names: Erectile Dysfunction
  Arms: Wait-list control

SUMMARY:
The investigators propose a single-site, prospective randomized trial to determine the effects of aerobic exercise training on ED among 50 sedentary men undergoing radical prostatectomy for clinically localized prostate cancer.

DETAILED DESCRIPTION:
We propose a single-site, prospective randomized trial to determine the effects of aerobic exercise training on ED among 50 sedentary men undergoing radical prostatectomy for clinically localized prostate cancer. This project has three specific aims:

* Specific Aim #1: To determine the effects of aerobic exercise training versus wait-list control on incidence of ED among sedentary men undergoing radical prostatectomy for clinically localized prostate cancer.
* Hypothesis #1: Aerobic exercise training will be associated with a significantly lower incidence of ED compared with usual care among sedentary men undergoing radical prostatectomy for clinically localized prostate cancer.
* Specific Aim #2: To determine the effects of aerobic exercise training versus wait-list control on changes in patient symptoms (i.e., erectile function score, sexual functioning, urinary incontinence, and QOL) and the number of men receiving phosphodiesterase type-5 (PDE-5) inhibitor therapy as well as therapy dose.
* Hypothesis #2: Aerobic exercise training will improve patient symptoms and reduce the number of men requiring PDE-5 inhibitor therapy.
* Specific Aim #3: To determine the effects of aerobic exercise training versus wait-list control on changes in postulated biologic mechanisms that may underlie the relationship between exercise training and ED [i.e., CVD risk factors (cardiorespiratory fitness, lipid profile, blood pressure, c-reactive protein, body composition), cardiac function, and penile and brachial artery endothelial function].
* Hypothesis #3: Aerobic exercise training will be associated with favorable changes in postulated candidate mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Legal age (>18 years old)
2. An interval of at least 4-6 weeks between prior radical prostatectomy and study enrollment. Radical prostatectomy-induced ED is an immediate and progressive disorder as such interventions shortly following surgery may be the most effective at attenuating this disorder. It is expected that men who have undergone radical prostatectomy will be fully recovered at 4-6 weeks post surgery and will be receptive to an exercise intervention study at this time (capitalizing on the teachable moment). Additionally, the PI has demonstrated that maximal cardiopulmonary exercise testing is a safe, feasible, and acceptable assessment procedure 7±3 days post-craniotomy among 20 primary high grade primary brain tumor patients and 30±5 days post-pneumonectomy or lobectomy among 20 operable non-small cell lung cancer patients,
3. Karnofsky performance status of at least 70% at study entry,
4. Estimated life expectancy of ≥6 months,
5. Ability to read and understand English,
6. Primary attending urologist approval (Drs. Donatucci and Moul),
7. Signed informed consent prior to initiation of study-related procedures,
8. Willingness to be randomized,
9. Sedentary (i.e., men not performing regular exercise on at least 5 days a week, for at least 30 minutes each session, at a moderate or vigorous intensity for the past month). This definition is consistent with the national exercise recommendations guidelines and will ensure that only men not currently engaging in regular exercise (i.e., those who are the most likely to benefit) are recruited,
10. Postoperative erectile function (score ≤21 on the International Index of Erectile Function (IIEF) multidimensional questionnaire90). To avoid potential ceiling effects (i.e., testing of the intervention among men with only good erectile function), only men with an IIEF score ≤21, which indicates ED, will be recruited.

Exclusion Criteria:

1. Presence of a concurrent, actively treated other malignancy or history of other malignancy treated within the past 3 years (other than non-melanoma skin cancer),
2. Presence of metastatic disease,
3. Scheduled to receive any form of adjuvant cancer therapy (i.e., radiation, chemotherapy, androgen deprivation therapy),
4. Subjects must not have any of following absolute contraindications to exercise testing as recommended by the American Thoracic Society91:

   * acute myocardial infarction (3-5 days)
   * unstable angina
   * uncontrolled arrhythmias causing symptoms or hemodynamic compromise
   * syncope
   * acute endocarditis
   * acute myocarditis or pericarditis
   * uncontrolled heart failure
   * acute pulmonary embolus or pulmonary infarction
   * thrombosis of lower extremities
   * suspected dissecting aneurysm
   * uncontrolled asthma
   * pulmonary edema
   * room air desaturation at rest ≤ 85%
   * respiratory failure
   * acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
   * mental impairment leading to inability to cooperate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the effects of supervised aerobic exercise training versus usual care on incidence of ED among men undergoing radical prostatectomy for clinically localized prostate cancer. | 12 months

SECONDARY OUTCOMES:
To determine the effects of aerobic exercise training versus wait-list control on changes in patient symptoms and the number of men receiving phosphodiesterases type-5 (PDE-5) inhibitor therapy as well as therapy dose. | 12 months
To determine the effects of aerobic exercise training versus wait-list control on changes in postulated biologic mechanisms that may underlie the relationship between exercise training and ED.
  To determine the effects of aerobic exercise training versus wait-list control on changes in postulated biologic mechanisms that may underlie the relationship between exercise training and ED [i.e., CVD risk factors (cardiorespiratory fitness, lipid profile, blood pressure, c-reactive protein, body composition), cardiac function, and penile and brachial artery endothelial function].

CONTACTS AND LOCATIONS:
Overall Officials: Lee W Jones, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States